CLINICAL TRIAL: NCT02724826
Title: Effects of Qigong and Exercise Therapy Among Patients With Chronic Neck Pain
Acronym: QII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Collaborators: Göteborg University (Other)
Responsible Party: Principal Investigator, Liselott Persson, RPT. PhD, Lund University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 516/99
Record Dates: First submitted 2016-03-07; First posted 2016-03-31 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Neck Pain
Keywords: Expectations; Outcomes; Qigong; Exercise therapy; Disability; Neck movements,
MeSH Terms: conditions — Neck Pain | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Qigong therapy (Experimental): The qigong treatment was done according to medical qigong, and is a way of affecting and directing qi (energy) for medical benefit. Each qigong practice included body posture adjustment, gentle movement, meditation, relaxation, breathing regulation practices and massage. The qigong was practiced in groups of ten to 15 participants. Each qigong session started with information about the philosophy and a general warm-up with soft movements and 14 selected qigong exercises according to the Biyun method.
  Interventions: Behavioral: Exercise therapy
- Exercise therapy (Active Comparator): Exercise therapy was carried out individually, adjusted for each participant. A physiotherapist instructed the participant with focused on the cervical and shoulder/thoracic regions. Each training session included stationary bicycle for ten minutes, 40 minutes of dynamic exercises. These exercises consisted of active movements in all neck directions and muscle exercises aimed to maintain/increase circulation, endurance and strength. The load at the muscle exercises was to achieve between 30 and 70% of maximum muscle capacity and was gradually increased as endurance and strength were gained.
  Interventions: Behavioral: Qigong therapy

INTERVENTIONS:
Behavioral: Qigong therapy — Medical qigong
  Arms: Exercise therapy
Behavioral: Exercise therapy — Regular exercise
  Arms: Qigong therapy

SUMMARY:
A randomized controlled, multicenter trial comparing qigong and exercise therapy concerning pain intensity, treatment expectations, disability, neck movements and quality of life in subjects with non-specific, long-term NP after three and twelve months.

DETAILED DESCRIPTION:
A randomized controlled, multicenter trial comparing qigong and exercise therapy concerning pain intensity, treatment expectations, disability, neck movements and quality of life in subjects with non-specific, long-term NP. A comparison will be performed between the two randomized treatment groups in these variables before and after three and 12 months.

Participants were recruited via an advertisement in a local newspaper. Inclusion: Men and women between 18-65 years of age with nonspecific, long term neck pain (<3 months).Exclusion criteria were chronic tension-type headache, migrain, traumatic neck injuries, neurologic signs or symptoms. rheumatic diseases, fibromyalgia or other severe physiologic or physical diserases and difficulties in understand the Swedish language.

The enrollment of participants, the randomization procedure and the performance of measurements were conducted by four independent physiotherapists. Randomization was done in blocks of 30 according to a sealed envelope technique. Assessments were made before treatment (baseline), immediately after treatment and at six and 12-month follow-ups. All participants answered questionnaires about demographic data, pain (duration and intensity) and disability. Pain intensity was rated as current NP and average NP during the week before the assessment, measured with a visual analogue scale (VAS - measured in millimeters with the end points 0 = no pain and 100 = unbearable pain) (Carlsson, 1983). Neck Movements was measured with cervico Thorac Ratio (CTR) (Norlander 2995), Disability was measured with the Neck Disability Index (NDI) (Vernon, 1991), which consists of a ten-item, scaled questionnaire where the total scores are recalculated into percent (0%, no disability; 100%, maximum disability). The items assess NP according to intensity, personal care, lifting, reading, headache, concentration, work, driving, sleeping and recreation. Quality of Life was measured with the SF-36 questionnaire (Sullivan1995).

Study participants One hundred and twenty-two subjects with long-term, non-specific NP were randomized to the interventions of qigong (n=60) and exercise therapy (n=62). Eighty-six (70%) were women and 36 (30%) men, with a mean age of 44 years

The participants were allocated randomly to receive qigong or exercise therapy. In each group, the participants received ten to 12 treatments over a period of three months, and each treatment session lasted one hour. A treatment-specific guideline was developed for each treatment. Treatments were provided by experienced physiotherapists; the physiotherapist responsible for qigong had nothing to do with exercise therapy and vice versa. An attendance list was kept during the intervention period, and all participants were informed that they had to attend at least eight of the 12 sessions to be included for analysis in the study.

Qigong was done according to medical qigong, which is a modality of traditional Chinese medicine and is a way of affecting and directing qi (energy) for medical benefit. There are several medical qigong techniques, one being the Biyun method . Each qigong practice included body posture adjustment and gentle movement, meditation (concentration) and purposeful relaxation, breathing regulation practices and self-administered massage. In this study, qigong was practiced in groups of ten to 15 participants. Each qigong session started with information about the philosophy of medical qigong, which was followed by a general warm-up with soft movements for the whole body and then 14 selected qigong exercises according to the Biyun method. The participants were recommended to practice different qigong exercises at home every day.

Exercise therapy was carried out individually, and the training program was adjusted for each participant. A physiotherapist instructed the participant throughout the training program, which focused mainly on the cervical and shoulder/thoracic regions. Each training session started with a warm-up on a stationary bicycle for about ten minutes, followed by 40 minutes of dynamic exercises. These exercises consisted of active movements aimed to cover the full range of motion in all neck directions and muscle exercises aimed to maintain/increase circulation, endurance and strength. The muscle exercises were carried out against gravity or with added resistance (for example with weights, rubber expander, dumbbells and pulley apparatus) and ended with stretching the muscles in the neck, shoulders and upper limbs. The amount of load was individualized and kept within pain tolerance (aimed not to increase pain). The load at the muscle exercises was to achieve between 30 and 70% of maximum muscle capacity and was gradually increased as endurance and strength were gained.

ELIGIBILITY:
Inclusion criteria:

* Men and women between 18-65 years of age
* nonspecific, long term neck pain (<3 months).

Exclusion criteria:

* chronic tension-type headache,
* migraine,
* traumatic neck injuries,
* neurologic signs or symptoms,
* rheumatic diseases,
* fibromyalgia or other severe physiologic or physical diseases
* difficulty in understand the Swedish language

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2000-08; Primary Completion 2004-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | 3 months and after 1 year
  measured with a visual analogue scale (VAS - measured in millimeters with the end points 0 = no pain and 100 = unbearable pain)

SECONDARY OUTCOMES:
Expectation | 3 months
  questionnaires
Disability, measured with the Neck Disability Index (NDI) | 3 months and after 1 year
  the Neck Disability Index (NDI) which consists of a ten-item, scaled questionnaire where the total scores are recalculated into percent (0%, no disability; 100%, maximum disability). The items assess NP according to intensity, personal care, lifting, reading, headache, concentration, work, driving, sleeping and recreation.
Quality of Life (SF36) | 3 months and after 1 year
  SF36 questionnaires consists of 36 statements subdivided into eight health-related dimensions: (1) physical functioning, (2) role physical: role limitations due to physical health problems, (3) bodily pain, (4) general health, (5) vitality: energy levels/fatigue, (6) social functioning, (7) role emotional: role limitations due to emotional problems, and (8) mental health: psychological distress Each scale has a maximum score of 100 and higher scores indicate higher subjective health.
Segmental flexion and mobility in the cervico-thoracic spine | 3 months and after 1 year
  assesssment with Myrin and Cervical Thoracal Ratio (CTR)

CONTACTS AND LOCATIONS:
Overall Officials: Lena-Karin Erlandsson, PhD, Study Chair — Head of Health Sciences Lund; Jane Y Carlsson, professor, Study Chair — Head of Health Sciences Gothenburg, jane.carlsson@neuro.gu.se

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Persson LCG, Lansinger B, Carlsson J, Gard G. Expectations of Qigong and Exercise Therapy in Patients With Long-term Neck Pain: An Analysis of a Prospective Randomized Study. J Manipulative Physiol Ther. 2017 Nov-Dec;40(9):676-684. doi: 10.1016/j.jmpt.2017.07.009. PMID 29229058
- Available data/document: Clinical Study Report — http://resolver.ebscohost.com/openurl?sid=Entrez%3aPubMed&id=pmid%3a18090079&site=ftf-live